CLINICAL TRIAL: NCT02681991
Title: Phase Ⅳ Clinical Trial to Evaluate of Renamezin in Patients With Chronic Renal Failure.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hyeong-Cheon Park, Principal Investigator, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNM-001
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

ARMS (1):
- test (Experimental): Renamezin capsule 2g, tid, PO
  Interventions: Drug: Renamezin capsule

INTERVENTIONS:
Drug: Renamezin capsule

SUMMARY:
Renamezin Capsule (an oral adsorbent) lowers indoxyl sulfate levels in patient with chronic renal failure.

120 patients with chronic renal failure(baseline serum creatinine:1.5-5.0mg/dl).

Renamezin is administered 6.0mg/day. The treatment period is 2 months. The change in serum indoxyl sulfate will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. patients spontaneously written consent to participate in this clinical trial
2. men and women over age of 19
3. pre-dialysis patients with chronic renal failure stage patient for 3 months and patients for holding the stable state in serum creatinine 1.5mg/dl - 5.0mg/dl
4. patients who were no noticeable change for 12weeks before screening and are expected to change is not needed during therapy in the therapy of chronic renal failure(medication and dose -related, diet therapy)

Exclusion Criteria:

1. patients with passes through the digestive tract disorders
2. patients with uncontrolled constipation symptoms
3. patients suffering from digestive tract ulcers and esophageal varices
4. patients with untreated severe hypertension (DBP ≥ 120mmHg)
5. patients hospitalized with angina pectoris, cardiovascular disease or diagnosed with serious arrhythmia or cerebrovascular disease within 6 months
6. patients with hepatic impairment (2 times greater than the upper limit of normal levels of AST, ALT)
7. subjects with dependency on alcohol
8. patients with current infections
9. pregnant women, nursing mothers
10. Patients with a possibility of pregnancy (However, negative case can be registered)
11. patients participating in another clinical trial in addition to the current clinical trial
12. Patient who do not fit the clinical trial participation the legal and mentally

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
change from baseline of Indoxyl sulfate at 8weeks | 0, 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Cheon Park, Professor, Principal Investigator — Gangnam Sevrance Hospital of Yonsei University
Locations (1):
- Gangnam Sevrance Hospital of Yonsei University, Seoul, Gangnam-gu, South Korea